CLINICAL TRIAL: NCT06635395
Title: Translation and Cross-Cultural Adaptation of the Baltimore Orthopedic Subscapularis Score Into Turkish
Brief Title: Turkish Validity and Reliability of Baltimore Orthopedic Subscapularis Score
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Research assistant, Istanbul Medeniyet University
Other Study IDs: BOSS
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Injuries; Subscapularis Tendon Tear
Keywords: scale validity; rotator cuff injuries; subscapularis tendon tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Rotator cuff injury: Scale validity and reliability The aim of this study is to adapt the Baltimore Orthopedic Subscapularis Score (BOSS) to Turkish society in patients with rotator cuff injury and to make its validity and reliability in Turkish. It has 5 questions. The patients will be sought to answer questionnaires during regular rehabilitation sessions.
  Interventions: Other: Scale validity and reliability

INTERVENTIONS:
Other: Scale validity and reliability — The aim of this study is to adapt the Baltimore Orthopedic Subscapularis Score (BOSS) to Turkish society in patients with rotator cuff injury and to make its validity and reliability in Turkish. It has 5 questions. The patients will be sought to answer questionnaires during regular rehabilitation sessions.

SUMMARY:
The aim of this study is to adapt the Baltimore Orthopedic Subscapularis Score (BOSS) to Turkish society and to make its validity and reliability in Turkish. The BOSS was developed by Hameker et al to differentiate subscapularis tears from other rotator cuff muscle tears in patients with rotator cuff injuries. The BOSS has 5 questions. This study will be conducted with patients with rotator cuff injuries. The patients will be sought to answer questionnaires during regular rehabilitation sessions. 25 participants will be included in the study. In order to evaluate the validity of the BOSS, the Western Ontario Rotator Cuff Disability Index (WORC), which can evaluate the functionality of the shoulder in patients with rotator cuff injury and has been validated in Turkish, and the SF-12 which can evaluate the quality of life and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

DETAILED DESCRIPTION:
The reliability and validity of the scale will begin with language equivalence and cultural adaptation. The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained from these two Turkish translations with a common opinion.

The scale, which has been translated into Turkish, will be translated into English by two other people who are fluent in Turkish and English. The scale translated into English will be compared with the original. In the pre-trial phase, a reassessment will be conducted with 15 participants to test the intelligibility of the scale. Based on the results of the pre-test phase, the final version of BOSS will be able to be modified. The data of BOSS will be collecting through face-to-face when the patients came to the rehabilitation center. 25 participants will be included in the study.

In order to evaluate the validity of the BOSS, the Western Ontario Rotator Cuff Disability Index (WORC), which can evaluate the functionality of shoulder in patients with rotator cuff injury and has been validated in Turkish, and the SF-12 which can evaluate the quality of life and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age who have been diagnosed with a rotator cuff injury,
* Patients whose native language is Turkish,
* Individuals with a Mini Mental State Examination score of >24,

Exclusion Criteria:

* Individuals with pain and disability due to any shoulder pathology other than rotator cuff injury,
* Individuals who cannot read or write Turkish,
* Individuals with shoulder fractures, surgical interventions and other accompanying shoulder pathologies,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with rotator cuff injury
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Disability | baseline
  Disability will be assessed with the Baltimore Orthopedic Subscapularis Score (BOSS) in patients with rotator cuff injuries. It has 5 items. Each item is scored on a 1-to-5, a total score ranging from 5 (best possible score) to 25 (worst possible score). Higher scores indicate a higher disability.
Functionality of the shoulder | baseline
  Functionality of the shoulder will be assessed with the Western Ontario Rotator Cuff Disability Index (WORC) in patients with rotator cuff injuries. It has 21 items. Each item is scored on a 0-to-100-mm visual analog scale, summing a total score ranging from 0 (best possible score) to 2100 (worst possible score). Higher scores indicate poorer functionality.

SECONDARY OUTCOMES:
Health status | baseline
  Health status will be assessed with the SF-12. It has 12 items. It has eight sub-dimensions and two summary scores: physical and mental. In the total score obtained from the scale, 100 indicates the best health status, while 0 indicates the worst health status.

CONTACTS AND LOCATIONS:
Overall Officials: emel mete, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No